CLINICAL TRIAL: NCT02342704
Title: A Multicenter, Randomized, Open-Label Study to Assess the Impact of Natalizumab Versus Fingolimod on Central Nervous System Tissue Damage and Recovery in Active Relapsing-Remitting Multiple Sclerosis Subjects
Brief Title: Impact of Natalizumab Versus Fingolimod in Relapsing-Remitting Multiple Sclerosis (RRMS) Participants
Acronym: REVEAL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101MS408; 2013-004622-29 (EudraCT Number)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab; Fingolimod Hydrochloride

ARMS (2):
- natalizumab (Experimental): Open-label natalizumab 300 mg IV every 4 weeks (Q4W)
  Interventions: Drug: natalizumab
- fingolimod (Active Comparator): Open-label fingolimod 0.5 mg once daily orally
  Interventions: Drug: fingolimod

INTERVENTIONS:
Drug: natalizumab — Administered as specified in the treatment arm
  Other Names: BG00002; Tysabri
  Arms: natalizumab
Drug: fingolimod — Administered as specified in the treatment arm
  Other Names: FTY720; Gilenya
  Arms: fingolimod

SUMMARY:
The primary objective of this study is to assess the effect of natalizumab compared to fingolimod on the evolution of new on-treatment T1-gadolinium-enhancing (Gd+) lesions to persistent black holes (PBH) over 52 weeks. The secondary objectives of this study in this study population are to assess the effect of natalizumab compared to fingolimod on: magnetic resonance imaging (MRI) measures of central nervous system (CNS) tissue destruction as measured by the number of new T1-Gd+ lesions; various other MRI measures of disease activity; No Evidence of Disease Activity (NEDA); Relapse on treatment over 52 weeks; The change in information processing speed as measured by the Symbol Digit Modalities Test (SDMT).

DETAILED DESCRIPTION:
This study also includes a Diffusion Tensor Imaging (DTI) sub-study that includes healthy volunteers. Healthy volunteers will not receive any study medication.

ELIGIBILITY:
Key Inclusion Criteria for MS Patients:

* Must have a documented diagnosis of relapsing MS (McDonald 2010 Criteria) at study screening with EDSS score from 0.0 to 5.5.
* If the subject is on Betaseron, Rebif, Avonex, Copaxone, Extavia, Tecfidera, and Aubagio (BRACE-TA) at study screening:
* He/she must have been on therapy for at least 6 months (unless experiencing highly active disease), have at least 9 T2-hyperintense lesions on a brain MRI scan, and have experienced ≥1 relapse within the last 6 months prior to study screening with ≥1 new T1-Gd+ lesion on a brain MRI scan performed ≤6 months prior to study screening or ≥2 new T2 lesions on a brain MRI scan performed ≤6 months prior to study screening, with comparison made to a T2 MRI scan performed up to 18 months before study screening
* If the subject has highly active disease, regardless of whether they are disease-modifying therapy (DMT)-naïve or had previous exposure to Betaseron, Rebif, Avonex, Copaxone, Extavia, Tecfidera, and Aubagio (BRACE-TA), they must have had ≥2 disabling relapses in the 12 months prior to study screening and either ≥1 new T1-Gd+ lesion on a brain MRI scan performed ≤6 months prior to study screening or ≥2 new T2 lesions on a brain MRI scan performed ≤6 months prior to study screening, with comparison made to a T2 MRI scan performed up to 18 months before study screening

Key Exclusion Criteria for MS Patients:

* Diagnosis of Primary Progressive Multiple Sclerosis and/or Secondary Progressive Multiple Sclerosis.
* History or positive test result at study screening for human immunodeficiency virus (HIV), hepatitis C virus (HCV) antibody or current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [HBcAb]).
* Prior treatment with natalizumab or fingolimod.
* History of or known active malignant disease, including solid tumors and hematologic malignancies (subjects with cutaneous basal and squamous cell carcinoma that has been completely excised and considered cured prior to study screening remain eligible).
* History of opportunistic infections or any clinically significant major disease, as determined by the Investigator.
* A clinically significant infectious illness (e.g., pneumonia, septicemia) within the 1 month prior to study screening.
* History of drug or alcohol abuse (as defined by the Investigator) within 1 year prior to study screening.
* Prior history of immunosuppressant use (e.g., mitoxantrone, azathioprine, methotrexate, cyclophosphamide, mycophenolate, cladribine, rituximab), or exposure to intravenous immunoglobulin (IGIV), monoclonal antibodies, cytokines, growth factors, soluble receptors, other recombinant products, or fusion proteins in the last 12 months prior to study screening.
* History of myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure in last 6 months.
* Treatment with Class Ia (e.g., procainamide, quinidine, ajmaline, disopyramide) or Class III (amiodarone, bretylium, dofelitide, sotalol, ibulitide, azilimide) anti-arrhythmic drugs.
* Concurrent therapy with drugs that slow heart rate (e.g., beta-blockers, heart-rate lowering calcium channel blockers such as diltiazem or verapamil, or digoxin).
* Hypertension not controlled with prescribed medications.
* History of severe respiratory disease, pulmonary fibrosis or class III or IV chronic obstructive pulmonary disease.
* The use of live or live attenuated vaccination within 8 weeks of study screening.

Key Inclusion Criteria for Healthy Volunteers:

* Subjects who are generally healthy as demonstrated by physical examination and by medical history, with no history or evidence of major illnesses, diseases, or disorders.
* Subjects of childbearing potential must practice effective contraception and be willing and able to continue contraception for duration of the study.
* No history of drug or alcohol abuse (as defined by the Investigator) within 1 year prior to study screening.

Key Exclusion Criteria for Healthy Volunteers:

* Claustrophobia sufficient to interfere with generating reliable MRI scans.
* History of other major illness including neurological disorders as determined by the Investigator.
* Presence of a metal device affected by MRI (e.g., any type of electronic, mechanical or magnetic implant, cardiac pacemaker, aneurysm clips, implanted cardiac defibrillator) or potential ferromagnetic foreign body (metal slivers, metal shavings, other metal objects), which would be a contraindication for MRI.
* Women who are currently pregnant or breastfeeding, or who have a positive pregnancy test result at screening.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2014-11-30 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2016-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (41):
- United States (12):
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Port Charlotte, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Des Moines, Iowa
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (3):
  - Research Site, Camperdown, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Heidelberg, Victoria
- Czechia (7):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Ostrava - Poruba
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Teplice
- France (3):
  - Research Site, Nîmes, Gard
  - Research Site, Libourne, Gironde
  - Research Site, Toulouse, Haute Garonne
- Germany (2):
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Erbach im Odenwald, Hesse
- Italy (2):
  - Research Site, Gianicolense, Roma
  - Research Site, Roma
- Spain (8):
  - Research Site, El Palmar, Murcia
  - Research Site, Málaga, Málaga
  - Research Site, Vigo, Pontevedra
  - Research Site, Santa Cruz de Tenerife, Tenerife
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Seville
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Stockholm
- United Kingdom (2):
  - Research Site, London, Greater London
  - Research Site, Glasgow, Strathclyde

REFERENCES:
- [Derived] Butzkueven H, Licata S, Jeffery D, Arnold DL, Filippi M, Geurts JJ, Santra S, Campbell N, Ho PR; REVEAL Investigators. Natalizumab versus fingolimod for patients with active relapsing-remitting multiple sclerosis: results from REVEAL, a prospective, randomised head-to-head study. BMJ Open. 2020 Oct 20;10(10):e038861. doi: 10.1136/bmjopen-2020-038861. PMID 33082194

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 128 participants were screened, 111 participants were enrolled in the study. Three participants were not randomized and did not receive any dose of study drug.
Groups:
- Natalizumab: Open-label natalizumab 300 mg IV every 4 weeks
Period: Overall Study
Arm/Group | Natalizumab | Fingolimod
Started | 54 (Safety Population: randomized participants who received at least 1 dose of study treatment.) | 54 (Safety Population: randomized participants who received at least 1 dose of study treatment.)
Completed | 1 | 3
Not Completed | 53 | 51
Not completed — Physician Decision | 0 | 3
Not completed — Sponsor Termination | 49 | 43
Not completed — Other | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natalizumab | Fingolimod | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.19 (8.811) | 34.87 (8.731) | 36.53 (8.887)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of ≥ 6-Month Confirmed T1-Hypointense Lesions Arising From New On-Treatment T1-Gadolinium-Enhancing (Gd+) Lesions
Time Frame: Up to Week 52
Population: The limited number of participants enrolled and the early termination of the study resulted in efficacy data not collected, and efficacy outcomes not analyzed, as per the pre-specified plan of analysis.
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cumulative Number of New T1-Gd+ Lesions
Time Frame: Baseline, Week 4, Week 12, Week 24
Population: Intent-to-treat population: all randomized participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 47 | 45
lesions
  From Baseline to Week 4 | 0.62 (1.512) | 1.69 (4.122)
  From Baseline to Week 12 | 0.68 (1.695) | 2.27 (4.499)
  From Baseline to Week 24 | 0.72 (1.69) | 2.6 (4.745)
Statistical Analysis 1: Comparison: Natalizumab vs Fingolimod; Week 4; Test type: Superiority or Other; p = 0.1260, Wilcoxon rank-sum test; p-value is based on Wilcoxon rank-sum test between the 2 treatment groups
Statistical Analysis 2: Comparison: Natalizumab vs Fingolimod; Week 4; Test type: Superiority or Other; p = 0.3525, negative binomial regression; p-value is based on negative binomial regression model, adjusted for baseline GD lesion count
Statistical Analysis 3: Comparison: Natalizumab vs Fingolimod; Week 12; Test type: Superiority or Other; p = 0.0127, Wilcoxon rank-sum test; p-value is based on Wilcoxon rank-sum test between the 2 treatment groups
Statistical Analysis 4: Comparison: Natalizumab vs Fingolimod; Week 12; Test type: Superiority or Other; p = 0.0299, negative binomial regression; p-value is based on negative binomial regression model, adjusted for baseline GD lesion count
Statistical Analysis 5: Comparison: Natalizumab vs Fingolimod; Week 24; Test type: Superiority or Other; p = 0.0123, Wilcoxon rank-sum test; p-value is based on Wilcoxon rank-sum test between the 2 treatment groups
Statistical Analysis 6: Comparison: Natalizumab vs Fingolimod; Week 24; Test type: Superiority or Other; p = 0.0076, negative binomial regression; p-value is based on negative binomial regression model, adjusted for baseline GD lesion count

3. Secondary Outcome: Change From Baseline in Total T1-Hypointense and Total T2-Hyperintense Lesion Volumes at Week 24
Description: As assessed by magnetic resonance imaging (MRI).
Time Frame: Baseline, Week 24
Population: Intent-to-treat population: all randomized participants who received at least 1 dose of study treatment and had an assessment.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 15 | 16
percentage change
  T1 Lesion Volume Change | 0.5 (31.235) | 1.81 (19.703)
  T2 Lesion Volume Change | 0.08 (4.399) | 3.32 (5.036)
Statistical Analysis 1: Comparison: Natalizumab vs Fingolimod; T1 Lesion Volume Change; Test type: Superiority or Other; p = 0.5318, Wilcoxon rank-sum test; p-value is based on Wilcoxon rank-sum test between the 2 treatment groups
Statistical Analysis 2: Comparison: Natalizumab vs Fingolimod; T2 Lesion Volume Change; Test type: Superiority or Other; p = 0.0528, Wilcoxon rank-sum test; p-value is based on Wilcoxon rank-sum test between the 2 treatment groups

4. Secondary Outcome: Change From Baseline in Total T1-Hypointense and Total T2-Hyperintense Lesion Volumes at Week 52
Description: As assessed by MRI.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 0 | 1
percentage change
  T1 Lesion Volume Change |  | -15.31 (NA) — only 1 participant had an assessment
  T2 Lesion Volume Change |  | 5.6 (NA) — only 1 participant had an assessment

5. Secondary Outcome: Cumulative Number of New or Enlarging T2 Lesions
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 15 | 16
lesions | 1.33 (2.469) | 1.94 (2.205)
Statistical Analysis 1: Comparison: Natalizumab vs Fingolimod; Test type: Superiority or Other; p = 0.2632, Wilcoxon rank-sum test; p-value is based on Wilcoxon rank-sum test between the 2 treatment groups

6. Secondary Outcome: Proportion of Participants With No Evidence of Disease Activity (NEDA)
Description: NEDA was defined as all of the following: no relapses; no 12-week confirmed disability progression based on Expanded Disability Status Scale (EDSS; defined as an increase of 1.0 or more on the EDSS from baseline of 1.0 or more, or an increase of 1.5 or more from a baseline score of 0) that was sustained for 12 weeks; no new T1-Gd+ lesions on brain MRI. No new or enlarging T2-hyperintense lesions.
Time Frame: Up to Week 52
Population: as for outcome 1
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to First Relapse
Description: A clinical relapse was defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement.
Time Frame: Up to Week 52
Population: as for outcome 1
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Cumulative Risk of Relapse
Description: as for outcome 7
Time Frame: Up to Week 52
Population: as for outcome 1
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Complete Recovery From First Relapse
Description: 12-week confirmed complete EDSS recovery from first on-treatment relapse is defined as an EDSS score that is equal to or lower than the last pre-relapse EDSS score and sustained for at least 12 weeks.
Time Frame: Up to Week 52
Population: as for outcome 1
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Symbol Digit Modalities Test (SDMT) at Week 24
Description: The SDMT measures the time to pair abstract symbols with specific numbers. The test requires elements of attention, visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items from 0-110 in 90 seconds. The total score provides a measure of the speed and accuracy of symbol-digit substitution.
Time Frame: Baseline, Week 24
Population: Intent-to-treat population: all randomized participants who received at least 1 dose of study treatment and had both baseline and post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 14 | 17
units on a scale | 3.79 (8.684) | 3.24 (4.63)

11. Secondary Outcome: Change From Baseline in SDMT at Week 52
Description: as for outcome 10
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Natalizumab | Fingolimod
Number analyzed (Participants) | 0 | 9
units on a scale |  | 2.11 (8.492)

ADVERSE EVENTS:
Time Frame: Up to 64 weeks.
Description: Treatment-emergent adverse events are presented.
Arm/Group | Natalizumab | Fingolimod
Serious Adverse Events (participants affected / at risk) | 0/54 | 2/54
Other Adverse Events (participants affected / at risk) | 14/54 | 23/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=54) | Fingolimod (N=54)
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=54) | Fingolimod (N=54)
Headache (Nervous system disorders) | 6 | 4
Multiple sclerosis relapse (Nervous system disorders) | 1 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 3
Migraine (Nervous system disorders) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 5
Urinary tract infection (Infections and infestations) | 2 | 3
Lymphocyte count decreased (Investigations) | 0 | 5
Alanine aminotransferase increased (Investigations) | 0 | 3
Anxiety (Psychiatric disorders) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Fatigue (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.